CLINICAL TRIAL: NCT00186693
Title: How Airway Remodeling and Hyperresponsiveness Contribute to Airflow Obstruction in Asthma
Status: Withdrawn | Type: Observational
Why Stopped: never received funding
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: GlaxoSmithKline (Industry)
Other Study IDs: 05-2453
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2006-07

CONDITIONS: Asthma
Keywords: Airway remodeling; Asthma; Hyper-responsiveness
MeSH Terms: conditions — Asthma; Airway Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Airway hyperresponsiveness is a characteristic feature of the asthma. It is known that there is an association between airway hyperresponsiveness and eosinophilic airway inflammation. However, even though inflammation can be reduced with appropriate asthma therapy, it is typical that airway hyperresponsiveness improves only modestly with treatment. The determinants of airway hyperresponsiveness are unclear.

It is also not clear as to the site of airway narrowing in asthma. It is hypothesized that airways beyond the 4th order have the greatest resistance.

We hope to determine the relationships between the airway inflammation, remodeling of the airway and airway hyperresponsiveness. Through local instillation of methacholine at bronchoscopy we will be able to study proximal and distal airways and the extent to which they constrict in vivo

DETAILED DESCRIPTION:
Airway hyperresponsiveness (AHR) is a characteristic feature of the asthmatic condition in humans. There is an association between AHR and eosinophilic airway inflammation. However, even though eosinophilic inflammation can be abolished with appropriate therapy, it is typical that AHR improves only modestly with treatment. The determinants of AHR are poorly understood. Recent data implicate mediators such as the cytokine Interleukin-13 (IL-13), structural changes to the airway wall (remodeling), increased contractility of airway smooth muscle cells (ASMC) and loss of mechanical connections or tethering, as potential factors contributing to AHR.

There is also uncertainty around the site of airway narrowing in asthma. In normal airways, bronchii around the 4th order have the greatest contribution to total resistance. It is hypothesized that the site of greatest resistance is moved distally in asthma and might even involve quite small airways close to the level of terminal bronchioles. Non-invasive methods to assess airway caliber in vivo are still unproven. One untested concern is that the airways of subjects with severe AHR have the potential to close completely putting them at risk of severe and even fatal airflow obstruction.

We propose to study AHR in humans with asthma: we will determine the relationships between AHR and (i) eosinophilic inflammation in the airway (sputum cellularity) via sputum induction, (ii) soluble mediators of inflammation (IL-13, IL-4, IL-5), (iii) remodeling of the airway wall (sub-epithelial fibrosis, ASMC accumulation)via biopsy. In addition we will compare measurements of AHR assessed by inhalation challenge with the results of direct, local installation of methacholine. At bronchoscopy, methacholine is delivered to the airway and bronchoconstriction is assessed directly. This method will allow study of proximal and distal airways, identification of heterogeneity of responses among airways and the extent to which human airways can constrict in vivo.

ELIGIBILITY:
Inclusion/ Exclusion Criteria:

* adults age 18 - 65 years
* stable asthma, defined as no need for new medical intervention in previous 4 weeks
* pre FEV1 > or = to 70% and able to have a methacholine challenge
* hyper-responsiveness as measured by methacholine challenge PC20 < or = 16 mg/ml
* steroid naive or stable inhaled corticosteroid medication in previous 8 weeks
* symptomatic treatment with bronchodilators permitted
* able to give written informed consent
* no other active/unstable medical conditions as judged by investigator
* subjects must be suitable for bronchoscopy in opinion of the investigator
* female subjects must no be pregnant, nursing or unwilling to use appropriate contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with asthma
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2006-09; Study Completion 2009-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Cox, MB FRCPC FRCPI, Principal Investigator — McMaster University
Locations (1):
- St Joseph's Healthcare, Hamilton, Ontario, Canada